CLINICAL TRIAL: NCT04598802
Title: A Physician-initiated, Multicentre, Ambispective, Observational Registry of Patients Undergoing Complex Aortic Procedures With the Use of the Bard Covera Plus (Tempe, Arizona, USA) Covered Self-expandable Stents
Brief Title: COvera in BRAnch Registry
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Bertoglio Luca, Principal Investigator, IRCCS San Raffaele
Other Study IDs: COBRA Registry
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Aneurysm
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covera Plus
  Interventions: Device: covered stent

INTERVENTIONS:
Device: covered stent — atherosclerotic aorto-iliac aneurysm

SUMMARY:
The purpose of the registry is to evaluate the peri-operative and short-, mid- and long-term outcomes of the Bard Covera Plus (Tempe, Arizona, USA) for the treatment of atherosclerotic aorto-iliac aneurysm in combination with a multibranched endograft

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥18 years
* Patients who underwent/will undergo a complex aortic procedure with the use of a Covera Plus covered stent graft as a bridging stent, in the centres involved in this Registry
* Subject has consented for study participation and signed the approved Informed Consent

Exclusion Criteria:

* Bleeding diathesis or coagulopathy
* Patients with active systemic or cutaneous infection or inflammation
* Patients who are pregnant or lactating
* Patient younger than 18 years of age
* Patients who did not receive treatment using a Covera Plus covered stent graft.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 patients treated from January 2018 to January 2022 for atherosclerotic aorto-iliac aneurysm with procedures requiring the use of the Covera Plus covered stent in combination with a branched endograft
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
technical success | 30 days
  freedom from type I or type III endoleak, stenosis/occlusion, dislocation/kinking
Branch instability | 30 days
  freedom from branch-related complications
Primary clinical success | 30 days
  freedom from death, type I/III endoleak, graft infection/thrombosis, aneurysm expansion and/or rupture, conversion to open repair, or new treatment-related thoraco-abdominal pathologies

CONTACTS AND LOCATIONS:
Locations (33):
- Germany (2):
  - University Heart & Vascular Center, Hamburg
  - Ludwig-Maximilians University Hospital, Munich
- Italy (31):
  - Ospedale di Asti, Asti
  - Ospedale Giuseppe Moscati, Avellino
  - Azienda Ospedaliero Universitaria Consorziale Policlinico, Bari
  - Fondazione Poliambulanza, Brescia
  - Azienda Ospedaliera di Cosenza, Cosenza
  - Azienda Ospedaliera Santa Croce e Carle, Cuneo
  - Ospedale civile San Giovanni di Dio, Florence
  - Ospedale Policlinico San Martino, Genova
  - Azienda Ospedaliera Universitaria Gaetano Martino, Messina
  - IRCCS San Raffaele, Milan
  - Ospedale Niguarda, Milan
  - Azienda Ospedaliera di Modena, Modena
  - Ospedale Cardarelli, Napoli
  - Azienda Ospedaliera di Padova, Padua
  - Ospedale Civico, Palermo
  - Azienda Ospedaliera Universitaria di Parma, Parma
  - Ospedale Pederzoli, Peschiera del Garda
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Ospedale San Camillo, Roma
  - Ospedale San Filippo Neri, Roma
  - Ospedale San Giovanni Addolorata Britannico, Roma
  - Policlinico Gemelli, Roma
  - Policlinico Umberto I, Roma
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Ospedale Molinette, Torino
  - Ospedale Santa Chiara, Trento
  - Ospedale Santa Maria di Ca' Foncello di Treviso, Treviso
  - Ospedale di Cattinara, Trieste
  - Azienda Ospedaliera di Verona, Verona
  - Ospedale Borgo Roma, Verona
  - Ospedale San Bortolo di Vicenza, Vicenza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mirza AK, Tenorio ER, Karkkainen JM, Hofer J, Macedo T, Cha S, Ozbek P, Oderich GS. Learning curve of fenestrated and branched endovascular aortic repair for pararenal and thoracoabdominal aneurysms. J Vasc Surg. 2020 Aug;72(2):423-434.e1. doi: 10.1016/j.jvs.2019.09.046. Epub 2020 Feb 17. PMID 32081482
- [Background] Tenorio ER, Oderich GS, Farber MA, Schneider DB, Timaran CH, Schanzer A, Beck AW, Motta F, Sweet MP; U.S. Fenestrated and Branched Aortic Research Consortium Investigators. Outcomes of endovascular repair of chronic postdissection compared with degenerative thoracoabdominal aortic aneurysms using fenestrated-branched stent grafts. J Vasc Surg. 2020 Sep;72(3):822-836.e9. doi: 10.1016/j.jvs.2019.10.091. Epub 2019 Dec 25. PMID 31882309
- [Background] Oikonomou K, Kopp R, Katsargyris A, Pfister K, Verhoeven EL, Kasprzak P. Outcomes of fenestrated/branched endografting in post-dissection thoracoabdominal aortic aneurysms. Eur J Vasc Endovasc Surg. 2014 Dec;48(6):641-8. doi: 10.1016/j.ejvs.2014.07.005. Epub 2014 Aug 28. PMID 25176618
- [Background] Verzini F, Parlani G, Varetto G, Gibello L, Boero M, Torsello GF, Donas KP, Simonte G; pELVIS Investigators. Late outcomes of different hypogastric stent grafts in aortoiliac endografting with iliac branch device: Results from the pELVIS Registry. J Vasc Surg. 2020 Aug;72(2):549-555.e1. doi: 10.1016/j.jvs.2019.09.065. Epub 2019 Dec 25. PMID 31882315
- [Background] Zhang J, Brier C, Parodi FE, Kuramochi Y, Lyden SP, Eagleton MJ. Incidence and management of iliac artery aneurysms associated with endovascular treatment of juxtarenal and thoracoabdominal aortic aneurysms. J Vasc Surg. 2020 Oct;72(4):1360-1366. doi: 10.1016/j.jvs.2019.12.040. Epub 2020 Mar 12. PMID 32173192
- [Background] Giosdekos A, Antonopoulos CN, Sfyroeras GS, Moulakakis KG, Tsilimparis N, Kakisis JD, Lazaris A, Chatziioannou A, Geroulakos G. The use of iliac branch devices for preservation of flow in internal iliac artery during endovascular aortic aneurysm repair. J Vasc Surg. 2020 Jun;71(6):2133-2144. doi: 10.1016/j.jvs.2019.10.087. Epub 2019 Dec 31. PMID 31901362
- [Derived] Bertoglio L, Grandi A, Veraldi GF, Pulli R, Antonello M, Bonvini S, Isernia G, Bellosta R, Buia F, Silingardi R; COBRA Registry Collaborators. Midterm results on a new self-expandable covered stent combined with branched stent grafts: Insights from a multicenter Italian registry. J Vasc Surg. 2023 Jun;77(6):1598-1606.e3. doi: 10.1016/j.jvs.2023.02.007. Epub 2023 Feb 22. PMID 36822256